CLINICAL TRIAL: NCT04650841
Title: The Role of the Opioid System in Placebo Effects on Pain and Social Rejection
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Responsible Party: Principal Investigator, Tor Wager, Diana L. Taylor Distinguished Professor, Trustees of Dartmouth College
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 230136
Record Dates: First submitted 2020-11-17; First posted 2020-12-03 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Pain; Rejection; Placebo Effect
MeSH Terms: conditions — Pain; Rejection, Psychology | interventions — Naloxone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Naloxone Group (Experimental): Participants will receive 4mg naloxone nasal spray.
  Interventions: Drug: Placebo Cream with Naloxone; Drug: Control Cream with Naloxone
- Saline Group (Experimental): Participants will receive saline in the nasal spray.
  Interventions: Drug: Placebo Cream with Saline; Drug: Control Cream with Saline

INTERVENTIONS:
Drug: Placebo Cream with Naloxone — Participants will be informed that the spray is an effective pain and negative emotion reducing agent.
  Arms: Naloxone Group
Drug: Control Cream with Naloxone — Participants will be informed that the spray is saline.
  Arms: Naloxone Group
Drug: Placebo Cream with Saline — Participants will be informed that the spray is an effective pain and negative emotion reducing agent.
  Arms: Saline Group
Drug: Control Cream with Saline — Participants will be informed that the spray is saline.
  Arms: Saline Group

SUMMARY:
The current study probes the involvement of the opioid system in placebo effects on social pain, using the opioid antagonist naloxone. 60 participants who recently experienced an unwanted breakup will experience rejection-related stimuli and receive painful heat and pressure stimuli during fMRI scanning. Participants will be randomized to receive either a naloxone or saline nasal spray, and be informed that the spray is either saline, or an effective pain and negative emotion reducing agent.

DETAILED DESCRIPTION:
Background:

Loss of close relationships is one of the most aversive life events. An unwanted romantic breakup leads to a 20% risk of developing depression within a month, a dramatic increase in depression risk. The investigators recently identified brain pathways mediating placebo effects on physical heat pain and the social pain associated with an unwanted breakup, including common involvement of dlPFC-PAG pathways and vmPFC. Other recent studies have identified rejection-related opioidergic activity in these circuits that may reflect endogenous regulatory mechanisms. This experiment probes the involvement of the opioid system in placebo effects on social pain, using the opioid antagonist naloxone.

Design:

Extending the investigator's previous design, participants who recently experienced an unwanted breakup will submit pictures of their ex-partners, places associated with strong memories of the partner, and written descriptions of memories that evoke rejection and social pain. Participants will 1) experience rejection-related stimuli and 2) receive painful heat and pressure stimuli in separate runs during fMRI scanning. FMRI scans after Control and Placebo treatment-nasal spray with suggestions of efficacy for emotion and pain-will be performed in a 2-session within-person counterbalanced design. Participants will be randomized into two groups that receive either (1) 4mg naloxone nasal spray or (2) saline in the nasal spray in both sessions, implementing a 2 x 2 (Placebo/Control x Saline/Naloxone) design.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-55 years
* No current psychiatric or major neurological diagnosis
* No reported substance abuse within the last six months
* Are capable of performing experimental tasks (e.g., are able to read, able to cooperate with fMRI examination)
* Are fluent or native speakers of English
* No current or recent history of pathological pain or reported neurological disorders.
* Having abstained from alcohol and substance use for 48 hours
* Passed fMRI safety screener
* Experienced a recent unwanted breakup of a romantic relationship

Exclusion Criteria:

* Current presence of pain
* Current or past history of primary psychiatric disorder
* Current or past history of psychoactive substance abuse or dependence
* Dementias
* Movement disorders except familial tremor
* CNS infection
* CNS vasculitis, inflammatory disease or autoimmune disease
* CNS demyelinating disease (e.g. multiple sclerosis)
* Space occupying lesions (mass lesions, tumors)
* Congenital CNS abnormality (e.g. cerebral palsy)
* Seizure disorder
* History of closed head trauma with loss of consciousness
* History of cerebrovascular disease (stroke, TIAs)
* Abnormal MRI (except changes accounted for by technical factors or UBOs)
* Neuroendocrine disorder (e.g., Cushings disease)
* Uncorrected hypothyroidism or hyperthyroidism
* Current or past history of cancer; Recent history (within two years) of myocardial infarction, severe cardiovascular disease, or currently active cardiovascular disease (e.g. angina, cardiomyopathy)
* Uncontrolled hypertension or hypotension
* Chronic pain syndromes
* Chronic fatigue syndromes
* Subjects unable to tolerate the scanning procedures (e.g., claustrophobia)
* Prior treatment within the last month with any of the following: antidepressants, mood stabilizers, glucocorticoids, opiates
* Prior treatment with any of the following: antipsychotics, isoniazid, centrally active antihypertensive drugs (e.g. clonidine, reserpine)
* Metal in body or prior history working with metal fragments (e.g., as a machinist)
* For women, pregnancy
* Any other contraindications for MRI examination (e.g., metallic implants such as pacemakers, surgical aneurysm clips, or known metal fragments embedded in the body)
* Claustrophobia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Intervention effects on pain ratings | Immediately after pain stimuli
  Pain ratings will be given on a 0-100 scale. 0 being "no pain at all" and 100 being "most pain imaginable in the context of this study."
Intervention effects on negative affect ratings | Immediately after rejection stimuli
  Rejection ratings will be given on a 0-100 scale. 0 being "not rejected at all" and 100 being "very rejected."
Brain: Pain signature response | Immediately after pain stimuli
  A priori regions of interest response from the brain (fMRI) patterns to the pain.
Brain: Rejection signature response | Immediately after rejection stimuli
  A priori regions of interest response from the brain (fMRI) patterns to rejection. The investigators will utilize a multivariate brain pattern developed and published in Woo et al., 2014, Nature Communications. This is a rejection-selected pattern of brain activity.
Skin conductance | Immediately after pain/rejection stimuli
  Skin conductance response (SCR) will be recorded during the task.
Heart rate | Immediately after pain/rejection stimuli
  Heart rate will be recorded during the task.

SECONDARY OUTCOMES:
Whole-brain maps of intervention effects | Immediately after pain/rejection stimuli
  Standard resting-state images will be acquired for exploratory analyses. Exploratory brain analysis will include univariate voxel-wise maps comparing participant groups with a threshold of q < 0.05, False Discovery Rate (FDR) corrected.
Rejection Sensitivity Questionnaire | Within 2 weeks before first fMRI scan
  A measure of sensitivity to actual or perceived rejection with ratings on a 6-point Likert scale ranging from "very unconcerned" - "very concerned." Higher scores indicate more reaction sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Tor D Wager, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth College, Hanover, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators are strongly committed to contributing to open and reproducible science. All MRI and behavioral data will be submitted to the NIMH Data Archive (NDA) according to the terms and conditions outlined on their website (https://ndar.nih.gov/contribute_data_sharing_regimen.html ) and with OpenFMRI.
  The investigators will ensure that our IRB has approved our Data Sharing Plan. The investigators will use an informed consent document that permits subjects to allow sharing of de-identified (face removed) MRI and fMRI data with open-sharing repositories, including the NDA and OpenFMRI databases. The consent form will stipulate that: "Scientists can use my information, without personal identifiers, for any kind of genetic research."
Time Frame: All data will be de-identified prior to sharing. Raw data will be submitted to NDA within one year from the end of data collection or 6 months from the acceptance date of the first primary study manuscript on the full dataset (excluding methods development papers), whichever is later. Analyzed data/maps of statistical results and models accompanying each paper will be submitted to NDA/OpenFMRI when the primary study manuscript is accepted.
Access Criteria: These data would generally be made available to any qualified investigator for neuroimaging studies only including:
  i. Research on any brain phenomenon; ii. Neuroimaging research on non-disease traits (intelligence, behavioral traits); iii. Methods development research.
  The requesting investigator must provide documentation of local IRB approval.
  These data would not be made available to:
  i. Any criminal justice organization, because data may not be used for any criminal justice applications; ii. Any commercial entity, because use of the data is limited to not-for-profit organizations and data may not be used for any commercial purposes.